CLINICAL TRIAL: NCT05628519
Title: Captain Sonar Impact on Trauma Patient Management
Acronym: CAST2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Claude Bernard University (Other)
Collaborators: Research on Healthcare Performance Lab U1290 (Other); Laboratoire Interuniversitaire de Biologie de la Motricité (Other)
Responsible Party: Principal Investigator, Lilot Marc, Clinical Professor, Claude Bernard University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: CAST2 N°20-119
Record Dates: First submitted 2022-05-18; First posted 2022-11-28 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Trauma Injury
Keywords: Healthcare professionals; Technical Skills; Non Technical Skills; Crew ressource Management; Stress evaluation and management
MeSH Terms: conditions — Accidental Injuries

STUDY DESIGN:
Intervention Model Description: Randomized control Trial, double blind
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Captain Sonar (Experimental): Participants will receive a training by a game session at Captain SonarTM of 60 min (including 15 min of presentation and prize in hand of the game) against a standardized investigator team
  Interventions: Behavioral: Captain Sonar Exposition
- Placebo Monopoly (Placebo Comparator): The control group participants will benefit from a 60 min session to play a "Placebo" game: monopoly
  Interventions: Behavioral: Monopoly Exposition

INTERVENTIONS:
Behavioral: Captain Sonar Exposition — Captain SonarTM is a naval battle game where two teams each composed of four participants clash. Each player has a well-defined role and it is imperative to communicate in a closed loop to advance in the game. This game also includes components similar to support for Trauma care: stress, speed of action, central communication and teamwork of four protagonists (Team Leader- Captain, intern-Second, nurse-Mechanic, Caregiver-Detector). This short video describes the rules and the Game progress: https://vimeo.com/173614346.
  Arms: Captain Sonar
Behavioral: Monopoly Exposition — Participant will be invited to play to Monopoly during 60 min
  Arms: Placebo Monopoly

SUMMARY:
Trauma patient care requires collaboration and interaction with close relationship between many stakeholders from different professions (senior doctor, intern, nurse, nurse helpers, surgeons, etc).

This is a stressful situation where decision and action need to be quick, decisive and coordinate.

In this situation, quality of care and patient safety depends on a good interprofessional communication.

The acquisition of advanced communication skills, team management and leadership, stress management are essentials elements in the practice of Intensive and trauma care. However, advanced structured training or assessment of theses skills is lacking in medical education or Healthcare professionals training. The study therefore, aimed to develop a global and attractive training to help healthcare professionals to improve their skills.

Captain SonarTM is a naval battle game where two teams each composed of four participants clash. Each player has a well-defined role and it is imperative to communicate in a closed loop to advance in the game. This game also includes components similar to support for shock management: stress, speed of action, central communication and teamwork of four protagonists (Team Leader-Captain, intern-Second, nurse-Mechanic, Nurse help-Detector). It may improve team building, team leadership, interprofessional work, communication, stress management. The study hypothesis is that this board game would have an impact on the performance of professionals when facing a multiple trauma simulated patient. (differences in terms of technical and non-technical performance. Different use of closed loop communication, Different stress management, different efficiency and interprofessional collaboration with potentially a reduction in the timing of treatment being delivered in trauma room)

DETAILED DESCRIPTION:
All the teams of 4 participants and 1 medical Student previously trained will then benefit from a training session either exposed to captain sonar or into the control arm with monopoly.

High-fidelity and multiprofessional simulation session based on the incoming of a severe traumatized patient will be held. These sessions will take place on high-fidelity mannequins lent by the CLESS (Lyonnais Center for Health Simulation Education) in pavilion H of Édouard Herriot Hospital, within the Trauma Center (in situ).

The same scenario will be presented for all groups (exposed and controls) with the same objectives of realization and the same complexity. An audio-visual recording will take place during each session in order to allow the evaluation of the study criteria on technical and non technical skills between the participants a posteriori of the simulation session.

ELIGIBILITY:
Inclusion Criteria:

Professional working at the Unit

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Technical skills | Measured during simulation session. Within 20 minutes of the simulation
  Total time of care in the trauma room, in seconds
Non technical skills | Measured during simulation session. Within 20 minutes of the simulation
  use of closed loop communications:
  - count of the number of closed loops/minute
Stress profile and stress management | immediately after simulation
  Visual Analog Scale of Stress, from 0 to 100 maximum

SECONDARY OUTCOMES:
Demographic data | At Baseline
  Demographic data (sex, age, previous experience as health care professional, experience in simulation, experience in gaming, experience in stress management)
Debriefing Evaluation | immediately After Debriefing
  Debriefing Assessment in Simulation in Healthcare (DASH) evaluated by team leader, nurse and facilitator, from 6 to 42 maximum
Influence of exposure on Performance, communication and stress management | immediately After simulation
  Visual analogic Scale, from 0 to 100 maximum
Technical skills grid | Measured during simulation session. Within 20 minutes of the simulation.
  Technical performance score (Grid out of 100 points); from 0 to 100 maximum
Technical skills key tasks | Measured during simulation session. Within 20 minutes of the simulation.
  Completion time for 5 key tasks (Hemocue result, blood pressure result, sample) in seconds Blood, realization of the FAST Ultrasound, Departure for OR/CT).
Technical skills self efficacy | Measured during simulation session. Within 20 minutes of the simulation.
  Self Efficacy estimation on Several cases, from 0 to 100 maximum Visual analog scale of support performance felt after the simulation session;
Non technical skills crew ressource 1 | Measured during simulation session. Within 20 minutes of the simulation.
  Non technical skills score : from 0 to 54 maximum
Non technical skills crew ressource 2 | Measured during simulation session. Within 20 minutes of the simulation.
  Non technical skills Score 2: from 1 to 5 maximum
Non technical skills communication anticipation | Measured during simulation session. Within 20 minutes of the simulation.
  Rate of anticipation of each participation (initiation of an act without prior request by the Team leader);
Non technical skills quality of team communication | immediately after simulation
  Visual Analog Scale quality of team communication, from 0 to 100 maximum.
Non technical skills confidence for team leader | immediately after simulation
  Visual Analog Scale of confidence in the team and the team leader , from 0 to 100 maximum.
Visual Analog Scale type of stress | immediately after the simulation session
  Visual Analog Scale of stress
Anxiety profile | immediately after the simulation session;
  Stait Trait Anxiety Inventory Trait, from 20 to 80 maximum.
Stress profiles and stress management physiological measurement heart rate variability | During Simulation within the 20 minutes of simulation
  Physiological stress assessment of 2 of each team members will be performed throughout inclusion (during exposure and during simulation) and measured by non-invasive and continuous recording:
  - Heart and respiratory rates and heart rate variability (Hexoskin® t-shirt)
Stress profiles and stress management electrodermal activity | During Simulation within the 20 minutes of simulation
  Electrodermal activity, reflecting the stress and activation of individuals (Empatica E4 watch on the wrist non-dominant)

CONTACTS AND LOCATIONS:
Locations (1):
- Anesthesiology and Intensive care medicine, H Building, Hopital Edouard Herriot, Hospices Civils de Lyon, Lyon, Rhone, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gawande AA, Zinner MJ, Studdert DM, Brennan TA. Analysis of errors reported by surgeons at three teaching hospitals. Surgery. 2003 Jun;133(6):614-21. doi: 10.1067/msy.2003.169. PMID 12796727
- [Background] Neily J, Mills PD, Young-Xu Y, Carney BT, West P, Berger DH, Mazzia LM, Paull DE, Bagian JP. Association between implementation of a medical team training program and surgical mortality. JAMA. 2010 Oct 20;304(15):1693-700. doi: 10.1001/jama.2010.1506. PMID 20959579
- [Background] El-Shafy IA, Delgado J, Akerman M, Bullaro F, Christopherson NAM, Prince JM. Closed-Loop Communication Improves Task Completion in Pediatric Trauma Resuscitation. J Surg Educ. 2018 Jan-Feb;75(1):58-64. doi: 10.1016/j.jsurg.2017.06.025. Epub 2017 Aug 2. PMID 28780315